CLINICAL TRIAL: NCT05351034
Title: The Role of High-resolution Anorectal Manometry in the Diagnosis of Functional Anorectal Disorders in Patients With Inactive Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Nader Ramzy Tamer, Assistant lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: HRAM in inactive IBD
Record Dates: First submitted 2022-04-02; First posted 2022-04-28 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Anorectal manometry — Anorectal manometry in diagnosis of Functional anorectal disorders

SUMMARY:
The study aimed at diagnose and to detect the incidence of functional anorectal disorders in patients with inactive inflammatory bowel disease and to highlight the role of anorectal manometry in evaluating IBD patients with persistent defecatory dysfunction .

DETAILED DESCRIPTION:
Inflammatory bowel diseases (IBD) are chronic disorders of the gastrointestinal tract associated with debilitating symptoms due to immune mediated enteric inflammation. Western countries have been historically observed that IBD is prevalent and continues to rise, whereas the general impression is that countries in the Middle East (ME) experience a lower incidence of IBD. Incidence rates vary considerably depending on the region. In 2017, Ulcerative Colitis (UC) incidence rates ranged from 0.97 to 57.9 per 100,000 in Europe, 8.8 to 23.14 per 100,000 in North America, and 0.15 to 6.5 per 100,000 in Asia and the ME. Nonetheless, recent trends have shown a significant rise in the incidence of IBD in Middle East countries, which were linked to "westernization" in lifestyle, including dietary habits in these countries .

Unfortunately IBD remains incurable .As a result, many patients experience intermittent flares of intestinal inflammation in an unpredictable relapsing-remitting pattern, with recognizable symptoms of increased bowel frequency, bleeding and urgency. While advances in the treatment of IBD in recent decades have increased the likelihood of achieving disease remission and mucosal healing, a significant proportion of patients still present with refractory gastrointestinal symptoms. In this context, there can be considerable overlap between symptoms in active IBD and overlapping coexisting functional gastrointestinal disorders in patients with quiescent disease.

Given the complexity of the normal continence and defecatory mechanism, it is unsurprising that disruption of one or more mechanism as a consequence of IBD can lead to either evacuatory dysfunction or fecal incontinence (FI) and multiple factors are involved in its pathogenesis.

Conventionally, Dyssynergic defecation ( DD) is an acquired behavioral disorder in which coordination is lacking between the pelvic floor/anal sphincter with abdominal muscles at the time of defecation. Among IBD patients, DD may be challenging to identify as it can present atypically with symptoms other than constipation, including urgency, rectal pain, sensation of incomplete evacuation, fecal incontinence, and frequent defecation.

This poses a significant challenge for clinicians, as failure to positively recognize functional disorders in patients without objective evidence of active inflammation, can lead to repeatedly negative and often invasive investigations, increased healthcare utilization, futile and potentially hazardous escalation of IBD therapies, and patient dissatisfaction due to refractory symptoms.

Anorectal manometry (ARM) is the most important test to assess anorectal function and detect motor abnormalities of sphincter function and anorectal coordination. It is indicated in patients presenting with FI and chronic refractory constipation and suspected evacuatory dysfunction. ARM enables assessment of rectal sensation,reflexes, and compliance. The manometric equipment will be used to measure the resting tone of the anal canal, voluntary function during squeeze, and reflex recto-anal coordination during rectal distension. In addition, it allows assessment for dyssynergic patterns and recto-anal coordination during simulated defecation ('push'). It is therefore a useful test to confirm physiological abnormalities to select patients for biofeedback therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older with IBD ,
* Patients have documented disease remission by endoscopy and laboratory data
* Patients have persistent defecatory symptoms .

Exclusion Criteria:

* Patients with a history of anorectal fistulizing / stricturing disease .
* Patients with prior surgery involving the anorectum .

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of functional anorectal disorders in patients with inactive inflammatory bowel disease with defecatory symptoms . | baseline
  To detect the possible association between inactive inflammatory bowel disease and functional anorectal disorders.

SECONDARY OUTCOMES:
Detect the average resting anal pressure among patients with inactive IBD | baseline
  using anorectal manometry to detect the anal canal pressure during rest
Detect the average anal pressure changes in respond to squeeze and cough among patients with inactive IBD | baseline
  using anorectal manometry to detect the anal canal pressure during coughing and squeezing
assess rectal sensation among patients with inactive IBD | baseline
  using anorectal manometry balloon insufflation to detect the rectal sensation pressure
Estimate recto-anal coordination in patients with inactive IBD | baseline
  using anorectal manometry to detect the coordination of anal sphincter in response to push
Estimate the anal sphincter inhibition in response to sudden change in rectal pressure ( RAIR ) in patients with inactive IBD | baseline
  Sudden insufflation of the balloon lead to reflex inhibition of internal anal sphincter in normal individuals .

REFERENCES:
- [Background] Sharara AI, Al Awadhi S, Alharbi O, Al Dhahab H, Mounir M, Salese L, Singh E, Sunna N, Tarcha N, Mosli M. Epidemiology, disease burden, and treatment challenges of ulcerative colitis in Africa and the Middle East. Expert Rev Gastroenterol Hepatol. 2018 Sep;12(9):883-897. doi: 10.1080/17474124.2018.1503052. Epub 2018 Aug 10. PMID 30096985
- [Background] Bryant RV, van Langenberg DR, Holtmann GJ, Andrews JM. Functional gastrointestinal disorders in inflammatory bowel disease: impact on quality of life and psychological status. J Gastroenterol Hepatol. 2011 May;26(5):916-23. doi: 10.1111/j.1440-1746.2011.06624.x. PMID 21214889
- [Background] Perera LP, Ananthakrishnan AN, Guilday C, Remshak K, Zadvornova Y, Naik AS, Stein DJ, Massey BT. Dyssynergic defecation: a treatable cause of persistent symptoms when inflammatory bowel disease is in remission. Dig Dis Sci. 2013 Dec;58(12):3600-5. doi: 10.1007/s10620-013-2850-3. Epub 2013 Sep 12. PMID 24026401
- [Background] Rao SS, Mudipalli RS, Stessman M, Zimmerman B. Investigation of the utility of colorectal function tests and Rome II criteria in dyssynergic defecation (Anismus). Neurogastroenterol Motil. 2004 Oct;16(5):589-96. doi: 10.1111/j.1365-2982.2004.00526.x. PMID 15500515
- [Background] Carrington EV, Scott SM, Bharucha A, Mion F, Remes-Troche JM, Malcolm A, Heinrich H, Fox M, Rao SS; International Anorectal Physiology Working Group and the International Working Group for Disorders of Gastrointestinal Motility and Function. Expert consensus document: Advances in the evaluation of anorectal function. Nat Rev Gastroenterol Hepatol. 2018 May;15(5):309-323. doi: 10.1038/nrgastro.2018.27. Epub 2018 Apr 11. PMID 29636555
- [Background] Scott SM, Carrington EV. The London Classification: Improving Characterization and Classification of Anorectal Function with Anorectal Manometry. Curr Gastroenterol Rep. 2020 Sep 15;22(11):55. doi: 10.1007/s11894-020-00793-z. PMID 32935278